CLINICAL TRIAL: NCT05518175
Title: Patient-centered Outcomes After Permanent Female Sterilization Procedure: A Randomized Controlled Trial Comparing Three Surgical Routes
Brief Title: Patient-centered Outcomes After Permanent Female Sterilization Procedure(POPS Trial)
Acronym: POPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Randa Jalloul, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-22-0470
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-06

CONDITIONS: Sterility, Female
Keywords: laparoscopy; quality of recovery; vaginal natural orifice transluminal endoscopic surgery
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Route A: Traditional laparoscopy (Active Comparator)
  Interventions: Procedure: Traditional laparoscopy
- Route B: Single site laparoscopy (Experimental)
  Interventions: Procedure: Single site laparoscopy
- Route C:V-Notes surgery (Experimental)
  Interventions: Procedure: V-Notes surgery

INTERVENTIONS:
Procedure: Traditional laparoscopy — Utilizes three or four ports for access and retrieval.
  Arms: Route A: Traditional laparoscopy
Procedure: Single site laparoscopy — One port is placed via a 2 to 3 cm umbilical/fascia incision. With this technique, there is a single incision, hidden in the umbilicus.
  Arms: Route B: Single site laparoscopy
Procedure: V-Notes surgery — One port placed trans-vaginally via a 2-3 cm vaginal incision with no abdominal scars.
  Arms: Route C:V-Notes surgery

SUMMARY:
The purpose of this study is to compare and capture key elements of the patient experience, quality of recovery, preferences and satisfaction after laparoscopic salpingectomy done via 3 different routes.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women scheduled to undergo an elective sterilization surgery regardless of parity
* non-prolapsed uterus
* Patients should able to provide written consent

Exclusion Criteria:

* Women who have relative contra-indication to vaginal peritoneal access such as: history of rectal surgery, suspected recto-vaginal endometriosis based on clinical history and examination, suspected malignancy, pelvic inflammatory disease, active lower genital tract infection, virginity or pregnancy
* Postpartum (immediate) tubal sterilization
* Tubal sterilization during a cesarean section

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Quality of recovery after surgery as assessed by the Quality of Recovery (QOR-40 )questionnaire | 24 hours after surgery
  This questionnaire has 40 questions, score varies from 40 (poor)-200 (excellent) a higher number indicating a better outcome

SECONDARY OUTCOMES:
Cosmesis as assessed by the Body Image Questionnaire | 2 weeks post surgery
  This includes 5 questions and each is scored on a 4-point Likert scale from 1(no, not at all) to 4(yes, extremely) with a maximum score of 20 and higher score indicating a better body image
Cosmesis as assessed by the Body Image Questionnaire | 6 weeks post surgery
  This includes 5 questions and each is scored on a 4-point Likert scale from 1(no, not at all) to 4(yes, extremely) with a maximum score of 20 and higher score indicating a better body image
Cosmesis as assessed by the Body Image Questionnaire | 3 months post surgery
  This includes 5 questions and each is scored on a 4-point Likert scale from 1(no, not at all) to 4(yes, extremely) with a maximum score of 20 and higher score indicating a better body image
Change in sexual function as assessed by the Short version of the Female Sexual Function Index (FSFI) | Baseline, 3 months post surgery
  This has 9 items that address sexual dysfunctions. Each of these items are scored on a six-point scale ranging from 0 to 5, higher the score the better sexual function.
Pain as assessed by the Resting Visual Analog Scale (VAS) | 24 hours post surgery
  Rating pain on a scale from 0 to 10, 0 is no pain and 10 is severe pain during a quiet breathing period (resting VAS)
Pain as assessed by the Resting Visual Analog Scale (VAS) | 2 weeks post surgery
  Rating pain on a scale from 0 to 10, 0 is no pain and 10 is severe pain during a quiet breathing period (resting VAS)
Pain as assessed by the Resting Visual Analog Scale (VAS) | 6 weeks post surgery
  Rating pain on a scale from 0 to 10, 0 is no pain and 10 is severe pain during a quiet breathing period (resting VAS)
Pain as assessed by the Resting Visual Analog Scale (VAS) | 3 months post surgery
  Rating pain on a scale from 0 to 10, 0 is no pain and 10 is severe pain during a quiet breathing period (resting VAS)
Pain as assessed by the Dynamic Visual Analog Scale (VAS) | 3 months post surgery
  Rating pain on a scale from 0 to 10, 0 is no pain and 10 is severe pain after a voluntary cough (dynamic VAS)
Patient satisfaction as assessed by the satisfaction scale | 3 months post surgery
  Patients will rate their satisfaction on a 5 point Likert scale from 1(very unsatisfied) to 5(very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Randa J Jalloul, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No